CLINICAL TRIAL: NCT03037944
Title: Levonorgestrel-releasing Intrauterine System Versus a Low-dose Combined Oral Contraceptive for Management of Adenomyosis Uteri
Acronym: LNG-IUDvsCOCs
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Asmaa Mamdoh Mohamdy, Researcher, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ASAD0316
Record Dates: First submitted 2016-07-10; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Adenomyosis
Keywords: Adenomyosis; Contraceptive pills; Levonorgestrel-releasing Intrauterine System
MeSH Terms: conditions — Adenomyosis | interventions — drospirenone and ethinyl estradiol combination; drospirenone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Group A-LNG (Experimental): The Levonorgestrel releasing intrauterine device - IUD- will be Metraplant-E, which is used in this study for group A, is a modified Levonorgestrel-releasing intrauterine system from the old IUD "Metraplant", Metraplant-E design has a T-shaped frame containing Levonorgestrel and Ethylene Vinyl Acetate as well as Barium Sulphate to make it radio-opaque, All the "T" frame, the bulb of 20 mm length and sleeves contain: Ethylene Vinyl Acetate, Levonorgestrel and Barium Sulphate, ensure more exposure of the endometrial surface to the system and hence expect more endometrial suppression.
  Interventions: Device: Metraplant-E
- Group B-COCs (Experimental): Group B will receive combined oral contraceptive pills (Yasmin) COCs which will be Monophasic pills that have a constant dose of both estrogen and progestins in each of the hormonal active pills throughout the entire cycle . Yasmin (ethinyl estradiol 0.03 mg/ drospirenone 3 mg) tablets, provides an oral contraceptive regimen, it will be used continuously for 6 months with stoppage after 3 months for withdrawal bleeding.
  Interventions: Drug: Yasmin

INTERVENTIONS:
Drug: Yasmin — (ethinyl estradiol 0.03 mg/ drospirenone 3 mg) tablets
  Other Names: drospirenone and ethinyl estradiol tablets
  Arms: Group B-COCs
Device: Metraplant-E — Levonorgestrel-releasing Intrauterine System modified levonorgestrel-releasing intrauterine system from the old IUD "Metraplant", modified by Azzam 2013
  Other Names: Metraplant-E- Levonorgestrel
  Arms: Group A-LNG

SUMMARY:
This study aims to compare the efficacy of LNG - IUD (Levonorgestrel releasing intrauterine device) Versus Low dose COCs (combined oral contraceptive pills) on management of heavy menstrual bleeding and Dysmenorrhea caused by Adenomyosis.

DETAILED DESCRIPTION:
Levonorgestrel releasing intrauterine device will be MetraPlant-E, which is used in this study in group A, is a modified Levonorgestrel -releasing intrauterine system from the old IUD - Intrauterine Device "Metraplant", MetraPlant-E design has a T-shaped frame containing Levonorgestrel and Ethylene Vinyl Acetate as well as Barium Sulphate to make it radio-opaque, All the "T" frame, the bulb of 20 mm length and sleeves contain: Ethylene Vinyl Acetate, Levonorgestrel and Barium Sulphate, which ensures more exposure of the endometrial surface to the system and hence expected more endometrial suppression.

It consists of Levonorgestrel Hormone (60 mg), Ethylene Vinyl Acetate (120 mg) & Barium Sulphate (20 mg) Metraplant-E is designed without any coat membrane, which will help in more rise in Levonorgestrel level (higher initial release). The high initial release of Levonorgestrel (reached more than 28µg/24hrs in Metraplant-E in this study of in-vitro release) may help in early stoppage of bleeding in patients who suffer from irregular bleeding.

Women in group A will receive IUD - Intrauterine Device- during menstruation .It will be inserted into uterus in similar procedure to non-hormonal IUD .Pelvic exam will be done, the vagina will hold open with speculum, grasping the cervix, measuring uterine length and proper insertion of IUD - Intrauterine Device by non-touch technic. Women will receive proper antibiotics after insertion.

Group B will receive combined oral contraceptive pills (Yasmin) which will be Monophasic pills have a constant dose of both estrogen and progestin in each of the hormonal active pills throughout the entire cycle . Yasmin (ethinyl estradiol 0.03 mg/ drospirenone 3 mg) tablets, it provides an oral contraceptive regimen, it will be used continuously for 6 months with stoppage after 3 months for withdrawal bleeding.

Both treatment arms (Metraplant E and Yasmin) will be followed up after 3 months and 6 month of patients' recruitment. Assessment of pain related symptoms will be done using visual analogue scale pain score, while assessment of menstrual improvement will be done using menstrual diary.

ELIGIBILITY:
Inclusion Criteria:

* Women patient aged 30-45 years
* Diagnosed adenomyosis by transvaginal ultrasound or MRI or 3D ultrasound
* Patient complains of heavy menstrual bleeding or dysmenorrhea or both
* Living in a nearby area to make follow-up reasonably possible
* Planning for birth spacing for at least 2 years.

Exclusion Criteria:

* Pregnancy or seeking fertility
* Severe underlying comorbidities (hepatic, oncological)
* Pelvic inflammatory disease
* Other cervical or uterine pathologies
* Deep venous thromboembolism
* Hormonal therapy contraindications
* Endometriosis or fibroid

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of pain by pain measurement score | 6 Months
  measurement of the pain score by questionnaire form filled by patients. this questionnaire is evaluated by numbers corresponding to each answer chosen by patients
Number of bleeding days | 6 Months
  number of bleeding days is reported by patients and compared to pre- treatment conditions to evaluate the bleeding painful process duration and whether the intervention treatment had any relieving effect

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Es Abbas, Lecturer, Principal Investigator — Ain Shams University - Maternity Hospital; Karim Mo Labib, Lecturer, Principal Investigator — Ain Shams University - Maternity Hospital; Karim AH Labib, Assistant, Study Chair — Ain Shams University - Maternity Hospital
Locations (1):
- Ain Shams University - Maternity Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Benagiano, G.; Brosens, I.; Habiba, M.